CLINICAL TRIAL: NCT01982747
Title: A Phase I, Placebo-Controlled, Double-Blind, 2-Period Crossover Study to Assess Cardiac and General Safety and Pharmacokinetics of a Single Subcutaneous Dose of 60 mg MGN1703 in Healthy Volunteers
Brief Title: A Phase I Study to Assess Cardiac and General Safety and Pharmacokinetics of 60 mg MGN1703
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mologen AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MGN1703-C04
Record Dates: First submitted 2013-11-06; First posted 2013-11-13 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: Healthy
Keywords: Cardiac Safety; General Safety; Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MGN - Placebo (Other): Subjects of the MGN-Placebo arm will receive 60mg MGN1703 as 2 s.c. injections of 2 ml each during period 1 and physiological saline solution as Placebo as 2 s.c. injections of 2 ml each during period 2
  Interventions: Drug: MGN-Placebo
- Placebo-MGN (Other): Subjects of the Placebo-MGN arm will receive physiological saline solution as Placebo as 2 s.c. injections of 2 ml each during period 1 and 60mg MGN1703 as 2 s.c. injections of 2 ml each during period 2
  Interventions: Drug: Placebo-MGN

INTERVENTIONS:
Drug: MGN-Placebo
  Arms: MGN - Placebo
Drug: Placebo-MGN
  Arms: Placebo-MGN

SUMMARY:
MGN1703 is being developed for use in treating cancerous tumors effecting the colon, skin, kidneys and lungs. The dosage form of MGN1703 under investigation is an injection.

The goal of this study is to evaluate the effects of MGN1703 on the electrical activity of the heart in healthy subjects and to look at general safety.

ELIGIBILITY:
Inclusion Criteria:

1. The subject signs an IRB/IEC-approved informed consent prior to any study-related procedures.
2. Subject is male or female with no less than 6 subjects per sex in the study.
3. Subject is 18 to 65 years of age.
4. Subject's BMI is ≤32 kg/m2.
5. Female subjects of childbearing potential must not be pregnant or lactating with a negative serum HCG pregnancy test result at Screening and a negative urine HCG pregnancy test result on Days -1 and 14 prior to receiving study medication.
6. Female subjects of childbearing potential and male subjects must use an adequate method of contraception from Screening until completion of the study. Acceptable methods of contraception are barrier methods (male condom, female condom, diaphragm, cervical cap, spermicide or IUD), surgical sterility (documented doctor's report of vasectomy, hysterectomy and/or bilateral oophorectomy) and/or postmenopausal status (defined as at least 1 year without menses as demonstrated by medical history or subject report).
7. Subject is in good health as determined by vital signs, medical history, physical exam, and safety laboratory analyses at Screening and during the study.

Exclusion Criteria:

1. Subject has used an investigational product within 30 days prior to screening or during the study.
2. Subject has used prescription or non-prescription drugs (including vitamins, minerals, and herbal/plant-derived preparations) within 2 weeks of Screening (excluding oral contraceptives, hormonal IUD, hormone replacement therapy and acetaminophen) unless deemed acceptable by the Investigator in consultation with the Sponsor.
3. Subject has a positive drug and/or alcohol test at Screening, Day -1 or Day 14.
4. The subject has a history of drug or alcohol abuse within 2 years before Screening.
5. The subject is unable to abstain from ingesting alcohol, caffeine, grapefruit or Grapefruit juice for 72 hour prior to dosing.
6. The subject has a clinically significant history of cardiovascular, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, and/or other major diseases or malignancy.
7. Subject has a history of cardiac disease or any risk factors for TdP including (but not limited to) unexplained syncope, cardiac arrest, unexplained cardiac arrhythmia, structural heart disease and family history of Long QT syndrome.
8. Subject has evidence of any of the following cardiac conduction abnormalities at Screening, Day -1 or Day 1 prior to receiving any study medication:

   1. QTcF interval >430 msec for males and >450 msec for females
   2. PR interval >240 msec or <110 msec
   3. Evidence of second- or third-degree AVB
   4. Electrocardiographic evidence of complete LBBB, complete RBBB or incomplete LBBB
   5. Intraventricular conduction delay with QRS duration >120 msec
   6. Heart rate <40 bpm or >90 bpm
   7. Pathological Q waves (defined as >40 msec or depth >0.4-0.5 mV)
   8. Evidence of ventricular pre-excitation
9. The safety laboratory analyses at Screening are outside the normal limits and considered by the Investigator as clinically significant.
10. Any acute or chronic condition that, in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in this clinical study, a history of noncompliance to medical regimens, or subjects who are considered to be potentially unreliable.

    1. The subject has a positive test result for HIV antibody.
    2. The subject has a positive test result for the hepatitis C antibody or the HBsAg.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
cardiac safety of MGN1703 as compared to placebo | within the first 5 days after dosing
  assessed by 12 lead ECG

SECONDARY OUTCOMES:
general safety of MGN1703 as compared to placebo | within 5 days after dosing
  assessed by the following measures: safety laboratory analysis, vital signs and physical examination

OTHER OUTCOMES:
PK parameters of MGN1703 | within 5 days after dosing
  assessed by the following measures: Cmax, tmax, t1/2, AUCτ

CONTACTS AND LOCATIONS:
Overall Officials: Carlos R Sanabria, MD, Principal Investigator — Spaulding Clinical
Locations (1):
- Spaulding Clinical, West Bend, Wisconsin, United States